CLINICAL TRIAL: NCT04613804
Title: Toripalimab as Maintenance Therapy in Patients With Driver-gene Negative Advanced NSCLC After First-line Chemotherapy ：a Single-arm Phase II Trial
Brief Title: Toripalimab as Maintenance Therapy in Patients With Driver-gene Negative Advanced NSCLC After First-line Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCOG001
Record Dates: First submitted 2020-09-05; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-09

CONDITIONS: NSCLC Stage IV
Keywords: driver-gene negative advanced NSCLC; maintenance treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — toripalimab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Intervention Model Description: This study is a single-center, single-arm Phase II study. Qualified subjects will be treated with toripalimab every three weeks as a treatment cycle. After every two cycles, they will be evaluated the efficacy of tumor treatment by imaging and the safety of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Toripalimab group (Experimental): Toripalimab 240mg ivgtt Q21d
  Interventions: Drug: Toripalimab Injection

INTERVENTIONS:
Drug: Toripalimab Injection — Qualified subjects will be treated with "toripalimab 240mg q21d" as a treatment cycle.
  Other Names: PD-1 inhibitor

SUMMARY:
Lung cancer is the malignant tumor with the highest incidence and mortality in China. Non-small cell lung cancer (NSCLC) ,which includes non-squamous cell carcinoma (including adenocarcinoma, large cell carcinoma, and other cell types) and squamous cell carcinoma, accounts for about 80% of lung cancer. Platinum-based two-drug chemotherapy is the first-line standard treatment for driver-gene negative advanced NSCLC, but most patients experience disease progression after 4 to 6 months. To extend the efficacy of first-line treatment, maintenance therapy is a logical clinical option for patients who are effective after 4 to 6 cycles of standard treatment. There is currently no standard regimen for maintenance treatment of NSCLC. We evaluated the effectiveness and safety of maintenance therapy with the anti-PD-1 monoclonal antibody (Toripalimab injection) followed by the first-line standard regimen in advanced NSCLC patients who are effective after standard treatment. With a view to exploring treatment methods that are effective for the maintenance treatment of driver-gene negative advanced NSCLC and have little toxic and side effects,thereby improving the survival prognosis of these patients.

DETAILED DESCRIPTION:
Platinum-based two-drug chemotherapy is the first-line standard treatment for driver-negative advanced NSCLC, but most patients experience disease progression after 4 to 6 months. To extend the efficacy of first-line treatment, maintenance therapy is a logical clinical option for patients who are effective after 4 to 6 cycles of standard treatment. There is currently no standard regimen for maintenance treatment of NSCLC. We evaluated the effectiveness and safety of the anti-PD-1 monoclonal antibody (Toripalimab injection) followed by maintenance therapy in advanced NSCLC that was effective in the first-line standard regimen.Thereby improving the survival prognosis of advanced NSCLC.

ELIGIBILITY:
Criteria:

Inclusion Criteria:

* Fully understand the research and voluntarily sign the informed consent form (ICF)
* Age 18 to 75 years
* Histological or cytological documentation of non-small cell lung cance.
* Diagnosed as stage IV by imaging (staging according to AJCC eighth edition).
* Gene test is negative for EGFR, ALK, ROS1 confirmed by molecular pathology (tissue, ARMS method or NGS).
* Previously received first-line standard chemotherapy for non-small cell lung cancer (platinum combined with third-generation chemotherapy drugs in a two-drug combination regimen: pemetrexed or paclitaxel or docetaxel or gemcitabine or vinorelbine combined with cisplatin or carboplatin), and which were assessed the effectiveness by imaging(SD, PR or CR).
* At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria measured within 4 weeks prior to registration.
* ECOG performance status 0-1
* Expected overall survival time≥3 months
* Adequate bone marrow, Coagulation function，hepatic and renal function should be assessed by the following laboratory requirements conducted within 7 days before starting study treatment:

  * Leukocytes ≥ 3.0 x109/ L, absolute neutrophil count (ANC) ≥ 1.5 x109/ L, platelet count ≥ 100 x109/ L, hemoglobin (Hb) ≥9g/ dL.
  * Total bilirubin ≤ 1.5 x the upper limit of normal (ULN).
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN.
  * Serum creatinine ≤ 1.5 x the ULN.
  * Calculated creatinine clearance or 24 hour creatinine clearance ≥ 40 mL/ min.
  * INR≤1.5, Activated partial thromboplastin time(APTT)≤1.5×ULN.
* Patients with hepatitis B virus (HBV) infection and inactive/asymptomatic HBV carriers, or patients with chronic or active HBV, if the HBV DNA is <500IU/ml, or 2500copies/ml at the time of screening,can enter the group.
* Male subjects and women of childbearing age must have contraception within 24 weeks from the start of the study to the last time of using the drug.

Exclusion Criteria:

* Tumor histology or cytology pathology confirmed with small cell lung cancer components or sarcomatoid lesions.
* Previously received any T-cell co-stimulation or immune checkpoint therapy, including but not limited to CTLA-4 inhibitors, PD-1 inhibitors, PD-L1 / 2 inhibitors or other drugs that target T cells.
* Major autoimmune diseases.
* Subjects who were vaccinated or planned to be vaccinated within 4 weeks before the first time using the study drug.
* LD, drug-induced pneumonia, radiation pneumonitis requiring steroid therapy, or clinically active pneumonia or severe pulmonary dysfunction.
* TB or subjects with a history of active tuberculosis infection ≤ 48 weeks before screening, whether or not treated.
* Symptomatic cardiac disease, such as: heart failure above NYHA level 2, unstable angina pectoris, myocardial infarction occurred within 24 weeks, clinically significant supraventricular or ventricular arrhythmias require treatment or intervention.
* Acquired immunosuppression (AIDS or major immunosuppressive agents)
* Suffering from active viral hepatitis. Defined as: Hepatitis B virus (HBV) infection and HBV DNA ≥ 2500 copies / ml; or Hepatitis C virus (HCV) infection (quantitative test results of anti-HCV positive and HCV RNA are greater than the lower limit of detection) .
* Mental illness, alcohol, drug or substance abuse
* Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 12 months
  PFS by investigator-reported measurements according to CT image. PFS was calculated from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.PD was defined as Overall Response by RECIST criteria v1.1 according to CT image.

SECONDARY OUTCOMES:
Overall survival time | Up to 36 months
  OS was calculated from the date of randomization to death from any cause.
Objective response rate | up to 12 months
  CR + PR rate according to the RECIST version 1.1 guidelines.
Disease control rate | up to 12 months
  CR + PR + SD rate according to the RECIST version 1.1 guidelines.
Adverse events rate | up to 12 months
  Adverse events were assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0.

OTHER OUTCOMES:
Changes in immune environment | up to 12 months
  Assess the expression of PD-1, PD-L1, and TILs in tumor tissues before and after first-line standard chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong He, master, Study Chair — Fujian Cancer Hospital
Locations (1):
- Fujian cancer hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No